CLINICAL TRIAL: NCT03075085
Title: Developing and Testing Implementation Strategies for Evidence-Based Obesity Prevention in Childcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 205335; K01DK110141-01 (NIH)
Record Dates: First submitted 2017-02-20; First posted 2017-03-09 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — SOSTDC1 protein, human

STUDY DESIGN:
Intervention Model Description: Investigators will use a Type 3 Hybrid Design to test the effectiveness of the enhanced implementation strategy (i.e., facilitation) on uptake while also assessing impacts of the intervention on child outcomes. Investigators expect that the effectiveness of WISE on child outcomes will vary by the level of implementation fidelity, and a Hybrid 3 design allows for us to explore this hypothesis. RE-AIM provides an evaluation framework to assess key aspects of intervention programs implemented in real-word settings. Investigators will modify and use The Organizational Readiness to Change Assessment (ORCA) as developed for use with the i-PARiHS framework to assesses change commitment (e.g., We value this change) and change efficacy (e.g., We can keep the momentum going) both prior to and during implementation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basic WISE strategy (Active Comparator): These participants will be asked to implement the basic WISE strategy used in previous studies.
  Interventions: Behavioral: WISE (We Inspire Smart Eating)
- Enhanced WISE strategy (Experimental): These participants will be asked to implement the enhanced WISE strategy.
  Interventions: Behavioral: WISE (We Inspire Smart Eating)

INTERVENTIONS:
Behavioral: WISE (We Inspire Smart Eating) — An enhanced implementation strategy for evidence-based obesity prevention in childcare

SUMMARY:
Investigators will pilot test the impact of an enhanced implementation strategy on implementation and child health outcomes using continuous formative evaluation. Investigators will test the hypothesis that better fidelity to the implementation strategy (WISE) is positively related to child outcomes (e.g., child fruit and vegetable intake, BMI).

DETAILED DESCRIPTION:
Investigators will determine whether the enhanced strategy is feasible, acceptable, and demonstrates improved implementation, fidelity, and sustainability using a Hybrid Type 3 implementation design. Investigators expect that the effectiveness of WISE on child outcomes will vary by the level of implementation fidelity, and a Hybrid 3 design allows for us to explore this hypothesis).

ELIGIBILITY:
Inclusion Criteria:

* Early childhood educators from our partnering Head Start agency

Exclusion Criteria:

* Secondary Outcome Inclusion Criteria:
* Children aged 3-5 years old in our partnering Head Start agency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 696 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taren M Swindle, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Juonala M, Magnussen CG, Berenson GS, Venn A, Burns TL, Sabin MA, Srinivasan SR, Daniels SR, Davis PH, Chen W, Sun C, Cheung M, Viikari JS, Dwyer T, Raitakari OT. Childhood adiposity, adult adiposity, and cardiovascular risk factors. N Engl J Med. 2011 Nov 17;365(20):1876-85. doi: 10.1056/NEJMoa1010112. PMID 22087679
- [Background] Pulgaron ER. Childhood obesity: a review of increased risk for physical and psychological comorbidities. Clin Ther. 2013 Jan;35(1):A18-32. doi: 10.1016/j.clinthera.2012.12.014. PMID 23328273
- [Background] Kalarchian MA, Marcus MD. Psychiatric comorbidity of childhood obesity. Int Rev Psychiatry. 2012 Jun;24(3):241-6. doi: 10.3109/09540261.2012.678818. PMID 22724645
- [Background] Gross RS, Mendelsohn AL, Fierman AH, Hauser NR, Messito MJ. Maternal infant feeding behaviors and disparities in early child obesity. Child Obes. 2014 Apr;10(2):145-52. doi: 10.1089/chi.2013.0140. Epub 2014 Mar 25. PMID 24665873
- [Background] Johnson SL, Bellows L, Beckstrom L, Anderson J. Evaluation of a social marketing campaign targeting preschool children. Am J Health Behav. 2007 Jan-Feb;31(1):44-55. doi: 10.5555/ajhb.2007.31.1.44. PMID 17181461
- [Background] Mennella JA. Ontogeny of taste preferences: basic biology and implications for health. Am J Clin Nutr. 2014 Mar;99(3):704S-11S. doi: 10.3945/ajcn.113.067694. Epub 2014 Jan 22. PMID 24452237
- [Background] Larson N, Ward DS, Neelon SB, Story M. What role can child-care settings play in obesity prevention? A review of the evidence and call for research efforts. J Am Diet Assoc. 2011 Sep;111(9):1343-62. doi: 10.1016/j.jada.2011.06.007. PMID 21872698
- [Background] Freedman MR, Alvarez KP. Early childhood feeding: assessing knowledge, attitude, and practices of multi-ethnic child-care providers. J Am Diet Assoc. 2010 Mar;110(3):447-51. doi: 10.1016/j.jada.2009.11.018. PMID 20184996
- [Background] Benjamin SE, Cradock A, Walker EM, Slining M, Gillman MW. Obesity prevention in child care: a review of U.S. state regulations. BMC Public Health. 2008 May 30;8:188. doi: 10.1186/1471-2458-8-188. PMID 18513424
- [Background] Sigman-Grant M, Christiansen E, Fernandez G, Fletcher J, Johnson SL, Branen L, Price BA. Child care provider training and a supportive feeding environment in child care settings in 4 states, 2003. Prev Chronic Dis. 2011 Sep;8(5):A113. Epub 2011 Aug 15. PMID 21843416
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Woolf SH, Johnson RE. The break-even point: when medical advances are less important than improving the fidelity with which they are delivered. Ann Fam Med. 2005 Nov-Dec;3(6):545-52. doi: 10.1370/afm.406. PMID 16338919
- [Background] Glasgow RE. What types of evidence are most needed to advance behavioral medicine? Ann Behav Med. 2008 Feb;35(1):19-25. doi: 10.1007/s12160-007-9008-5. Epub 2008 Feb 12. PMID 18347901
- [Background] Clarke AM, Bunting B, Barry MM. Evaluating the implementation of a school-based emotional well-being programme: a cluster randomized controlled trial of Zippy's Friends for children in disadvantaged primary schools. Health Educ Res. 2014 Oct;29(5):786-98. doi: 10.1093/her/cyu047. Epub 2014 Aug 11. PMID 25113283
- [Background] Atkins MS, Frazier SL, Leathers SJ, Graczyk PA, Talbott E, Jakobsons L, Adil JA, Marinez-Lora A, Demirtas H, Gibbons RB, Bell CC. Teacher key opinion leaders and mental health consultation in low-income urban schools. J Consult Clin Psychol. 2008 Oct;76(5):905-8. doi: 10.1037/a0013036. PMID 18837608
- [Background] Eiraldi R, McCurdy B, Khanna M, Mautone J, Jawad AF, Power T, Cidav Z, Cacia J, Sugai G. A cluster randomized trial to evaluate external support for the implementation of positive behavioral interventions and supports by school personnel. Implement Sci. 2014 Jan 15;9:12. doi: 10.1186/1748-5908-9-12. PMID 24428904
- [Background] Noell GH, Witt JC, LaFleur LH, Mortenson BP, Ranier DD, LeVelle J. Increasing intervention implementation in general education following consultation: a comparison of two follow-up strategies. J Appl Behav Anal. 2000 Fall;33(3):271-84. doi: 10.1901/jaba.2000.33-271. PMID 11051568
- [Background] Rabin BA, Glasgow RE, Kerner JF, Klump MP, Brownson RC. Dissemination and implementation research on community-based cancer prevention: a systematic review. Am J Prev Med. 2010 Apr;38(4):443-56. doi: 10.1016/j.amepre.2009.12.035. PMID 20307814
- [Background] Bell AC, Davies L, Finch M, Wolfenden L, Francis JL, Sutherland R, Wiggers J. An implementation intervention to encourage healthy eating in centre-based child-care services: impact of the Good for Kids Good for Life programme. Public Health Nutr. 2015 Jun;18(9):1610-9. doi: 10.1017/S1368980013003364. Epub 2014 Jan 9. PMID 24477181
- [Background] Jones J, Wolfenden L, Wyse R, Finch M, Yoong SL, Dodds P, Pond N, Gillham K, Freund M, McElduff P, Wye P, Wiggers J. A randomised controlled trial of an intervention to facilitate the implementation of healthy eating and physical activity policies and practices in childcare services. BMJ Open. 2014 Apr 17;4(4):e005312. doi: 10.1136/bmjopen-2014-005312. PMID 24742978
- [Background] Ermakov IV, Gellermann W. Dermal carotenoid measurements via pressure mediated reflection spectroscopy. J Biophotonics. 2012 Jul;5(7):559-70. doi: 10.1002/jbio.201100122. Epub 2012 Feb 13. PMID 22331637
- [Background] Scarmo S, Henebery K, Peracchio H, Cartmel B, Lin H, Ermakov IV, Gellermann W, Bernstein PS, Duffy VB, Mayne ST. Skin carotenoid status measured by resonance Raman spectroscopy as a biomarker of fruit and vegetable intake in preschool children. Eur J Clin Nutr. 2012 May;66(5):555-60. doi: 10.1038/ejcn.2012.31. Epub 2012 Mar 21. PMID 22434053
- [Background] Khoo HE, Prasad KN, Kong KW, Jiang Y, Ismail A. Carotenoids and their isomers: color pigments in fruits and vegetables. Molecules. 2011 Feb 18;16(2):1710-38. doi: 10.3390/molecules16021710. PMID 21336241
- [Background] Darvin ME, Fluhr JW, Caspers P, van der Pool A, Richter H, Patzelt A, Sterry W, Lademann J. In vivo distribution of carotenoids in different anatomical locations of human skin: comparative assessment with two different Raman spectroscopy methods. Exp Dermatol. 2009 Dec;18(12):1060-3. doi: 10.1111/j.1600-0625.2009.00946.x. PMID 19650865
- [Background] Blume-Peytavi U, Rolland A, Darvin ME, Constable A, Pineau I, Voit C, Zappel K, Schafer-Hesterberg G, Meinke M, Clavez RL, Sterry W, Lademann J. Cutaneous lycopene and beta-carotene levels measured by resonance Raman spectroscopy: high reliability and sensitivity to oral lactolycopene deprivation and supplementation. Eur J Pharm Biopharm. 2009 Sep;73(1):187-94. doi: 10.1016/j.ejpb.2009.04.017. Epub 2009 May 13. PMID 19442725
- [Background] Meinke MC, Darvin ME, Vollert H, Lademann J. Bioavailability of natural carotenoids in human skin compared to blood. Eur J Pharm Biopharm. 2010 Oct;76(2):269-74. doi: 10.1016/j.ejpb.2010.06.004. Epub 2010 Jun 15. PMID 20558286
- [Background] Levi J, Segal L, St. Laurent R, Rayburn J. The state of obesity: Better policies for a healthier America. Princeton (NJ): Robert Wood Johnson Foundation and Trust for America's Health; 2014 Sept. Available from: http://www.rwjf.org/en/library/research/2014/09/the-state-of-obesity.html
- [Background] Segal LM, Rayburn J, Martin A. Adult Obesity in the United States. Princeton (NJ): Robert Wood Johnson Foundation and Trust for America's Health; 2015. Available from: http://stateofobesity.org/adult-obesity/
- [Background] Frisvold DE, Lumeng JC. Expanding exposure: Can increasing the daily duration of head start reduce childhood obesity? The Journal of Human Resources 46(2): 373-402, 2011.
- [Background] Faith MS, Pietrobelli A, Heo M, Johnson SL, Keller KL, Heymsfield SB, Allison DB. A twin study of self-regulatory eating in early childhood: estimates of genetic and environmental influence, and measurement considerations. Int J Obes (Lond). 2012 Jul;36(7):931-7. doi: 10.1038/ijo.2011.258. Epub 2012 Jan 17. PMID 22249227
- [Background] Thomsen MR, Nayga RM, Alviola PA, Rouse HL. The effect of food deserts on the body mass index of elementary school children. American Journal of Agricultural Economics 98(1): 1-18, 2015.
- [Background] Dev DA, Speirs KE, McBride BA, Donovan SM, Chapman-Novakofski K. Head Start and child care providers' motivators, barriers and facilitators to practicing family-style meal service. Early Childhood Research Quarterly 29(4): 649-659, 2014.
- [Background] Child Care Aware of America. Child care in America: 2012 state fact sheets; 2012. Available from: http://usa.childcareaware.org/advocacy-public-policy/resources/reports-and-research/
- [Background] Whiteside-Mansell L, Bradley R, Conners N, Bokony P. The family map: Structured family interview to identify risks and strength in Head Start families. NHSA Dialog 10(3-4): 189-209, 2007.
- [Background] Darvin ME, Sterry W, Lademann J, Vergou T. The role of carotenoids in human skin. Molecules 16(12): 10491-10506, 2011.
- [Background] Darvin ME, Gersonde I, Meinke M, Sterry W, Lademann J. Non-invasive in vivo determination of the carotenoids beta-carotene and lycopene concentrations in the human skin using the Raman spectroscopic method. Journal of Physics D: Applied Physics 38(15): 2696, 2005.
- [Derived] Swindle T, McBride NM, Selig JP, Johnson SL, Whiteside-Mansell L, Martin J, Staley A, Curran GM. Stakeholder selected strategies for obesity prevention in childcare: results from a small-scale cluster randomized hybrid type III trial. Implement Sci. 2021 May 1;16(1):48. doi: 10.1186/s13012-021-01119-x. PMID 33933130
- [Derived] Swindle T, Selig JP, Rutledge JM, Whiteside-Mansell L, Curran G. Fidelity monitoring in complex interventions: a case study of the WISE intervention. Arch Public Health. 2018 Aug 29;76:53. doi: 10.1186/s13690-018-0292-2. eCollection 2018. PMID 30181874
- [Derived] Swindle T, Johnson SL, Whiteside-Mansell L, Curran GM. A mixed methods protocol for developing and testing implementation strategies for evidence-based obesity prevention in childcare: a cluster randomized hybrid type III trial. Implement Sci. 2017 Jul 18;12(1):90. doi: 10.1186/s13012-017-0624-6. PMID 28720140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 771 individuals were included in all study activities/aims. 488 individuals were included in the study trial.
Units Other Than Participants: Childcare centers
Groups:
- Basic WISE Strategy: These participants were asked to implement WISE using a basic implementation strategy (training and reminders only)
- Enhanced WISE Strategy: These participants were asked to implement WISE and supported with an Enhanced multi-faceted implementation strategy including a leadership commitment, an implementation blueprint, a local champion, an environmental reminder of the EBPs, facilitation, and tailored educational resources and incentives.
Period: Overall Study
Arm/Group | Basic WISE Strategy | Enhanced WISE Strategy
Started | 352; 5 Childcare centers | 344; 4 Childcare centers
Completed | 247; 5 Childcare centers | 232; 4 Childcare centers
Not Completed | 105; 0 Childcare centers | 112; 0 Childcare centers

BASELINE CHARACTERISTICS:
Population: At baseline, the Basic WISE strategy included 210 children and 36 teachers. At baseline, the Enhanced WISE strategy included 203 children and 39 teachers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Basic WISE Strategy | Enhanced WISE Strategy | Total
Number analyzed (Participants) | 246 | 242 | 488
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 210 | 203 | 413
  Between 18 and 65 years | 30 | 31 | 61
  >=65 years | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] — This refers to the age of the child. Age of teacher was collected categorically without measures of dispersion. Population: This refers to age of the child. Age of teacher was collected categorically.
  years
    number analyzed (Participants) | 210 | 203 | 413
    (all) | 4.1 (0.6) | 4.1 (0.6) | 4.1 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 147 | 315
  Male | 78 | 95 | 173
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 152 | 186 | 338
  White | 32 | 36 | 68
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 55 | 16 | 71
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 246 | 242 | 488
Carotenoid Intake [Mean (Standard Deviation); unit: resonance raman spectroscopy units] — This is a baseline measure for children in the study only, not teachers Population: This is a baseline measure for the children in the study only.
  resonance raman spectroscopy units
    number analyzed (Participants) | 210 | 203 | 413
    (all) | 25403.9 (9032.6) | 24732.8 (9041.3) | 25340.6 (9031.98)

OUTCOME MEASURES:

1. Primary Outcome: Change in Educators' Observed Implementation Fidelity Scores for Use of Evidence-Based Obesity Practices
Description: The WISE fidelity measure will be used across the school year. The WISE fidelity instrument is rated on a 1 to 4 scale with 4 representing the highest level of fidelity. Each core component is assessed with 2 items. Average fidelity scores above 3 are considered to reflect adequate fidelity on a component. That is, the 2 items on each fidelity component were averaged; an average of above 3 was considered as having achieved fidelity. We are reporting on the total number of classrooms that achieved fidelity in each condition at the spring (final assessment) for the evidence-based practices of WISE.
Time Frame: From Baseline Up to 8 months
Population: This measure is at the classroom level. Since there are 2 teachers per classroom, the number of classrooms is 18 and 19, respectively. That is, only one teachers per classroom provided data on this outcome. There are multiple classrooms per site, ranging from 1 to 6.
Measure: Count of Units; unit: Classrooms
Units Other Than Participants: Classrooms
Groups:
- Basic WISE Strategy: These classrooms were asked to implement WISE using a basic implementation strategy (training and reminders only).
- Enhanced WISE Strategy: These classrooms were asked to implement WISE and supported with an Enhanced multi-faceted implementation strategy including a leadership commitment, an implementation blueprint, a local champion, an environmental reminder of the EBPs, facilitation, and tailored educational resources and incentives.
Arm/Group | Basic WISE Strategy | Enhanced WISE Strategy
Number analyzed (Participants) | 18 | 19
Number analyzed (Classrooms) | 18 | 19
Classrooms
  Role Modeling | 4 | 10
  Use of Mascot | 2 | 4
  Hands On Exposure | 1 | 6

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 9 months from enrollment
Description: Through study completion, an average of 9 months from enrollment
Arm/Group | Basic WISE Strategy | Enhanced WISE Strategy
All-Cause Mortality (participants affected / at risk) | 0/352 | 0/344
Serious Adverse Events (participants affected / at risk) | 0/352 | 0/344
Other Adverse Events (participants affected / at risk) | 0/352 | 0/344

LIMITATIONS AND CAVEATS:
The turnover documented in this study (43% of teacher positions overall) is notably higher than national estimates for Head Start turnover (17-20%). Further, the uncertainty of the program's funding and the news of coming layoffs and site/classroom moves near the end of the trial were disruptive. The research team adapted to these changes in delivery of implementation strategies (e.g., facilitation to new educators) and data interpretation (i.e., focus on univariate analyses).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT03075085/Prot_SAP_000.pdf